CLINICAL TRIAL: NCT00794781
Title: A Phase 1, Multicenter, Open-Label, Dose-Escalation, Safety, Pharmacokinetic, and Pharmacodynamic Study of E6201 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E6201-A001-102
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Advanced Solid Tumors
Keywords: Cancer; solid tumors
MeSH Terms: conditions — Neoplasms | interventions — 14-(ethylamino)-8,9,16-trihydroxy-3,4-dimethyl-3,4,9,19-tetrahydro-1H-2-benzoxacyclotetradecine-1,7(8H)-dione

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E6201

INTERVENTIONS:
Drug: E6201 — E6201 Part A (Dose Escalation): Intravenous (IV) infusion administered over 30 minutes once weekly for 3 weeks (Days 1, 8, and 15). The first 3 to 6 subjects of the first cohort will receive 20 mg/m^2/week for a cycle of 3 weeks followed by a 1-week rest period. Subsequent dose escalations may increase at increments of 100% until two Grade 2 toxicities or 1 dose-limiting toxicity (DLT) are observed in a dose group. Thereafter, doses will be increased in increments of 50% or less until the maximum tolerated dose (MTD) is determined. Part B (MTD Expansion): After the MTD is determined in Part A, 15 additional subjects will continue to receive cycles at the MTD.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD), safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary anti-tumor activity of E6201 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible to participate in this study:

1. Willing and able to comply with the protocol and provide written informed consent.
2. Age greater than or equal to 18 years.
3. Histologically and/or cytologically confirmed metastatic melanoma which has progressed after treatment with approved therapies or for which there are no standard effective therapies available. CNS metastases from a primary melanoma are allowed.
4. Subjects must have melanoma tumor status established by a BRAF-gene analysis report from a CLIA qualified laboratory.
5. Subjects must have at least one tumor lesion accessible to biopsy in addition to one which is accurately and serially measurable according to RECIST 1.0 using either CT/MRI or photography (as appropriate), and which measures greater than 1.5 cm in the longest diameter for a non-lymph node and greater than 2.0 cm in the short axis diameter for a lymph node.
6. Female subjects of childbearing potential must agree to use medically acceptable methods of contraception, such as abstinence, double-barrier method (e.g., condom and spermicide; condom, diaphragm, and spermicide), intrauterine device (IUD), or have a vasectomised partner. Female subjects who use hormonal contraceptives must also use an additional approved method of contraception (as described previously). Contraceptive measures must start either prior to or at Screening and continue throughout the entire study period and for 2 months after the last dose drug is administered. Pregnant and/or lactating females are excluded.
7. Male subjects must agree to use contraceptive methods such as abstinence, or double-barrier method (e.g., condom and spermicide; condom, diaphragm, and spermicide). Contraceptive measures must start either prior to or at Screening and continue throughout the entire study period and for 2 months after the last dose of study drug is administered.
8. Adequate bone marrow function defined as:

   * Absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9/L
   * Hemoglobin greater than or equal to 9.0 g/dL; however, a hemoglobin value less than 9.0 g/dL is acceptable if it is corrected to greater than or equal to 9.0 g/dL by growth factor or transfusion before the start of treatment
   * Platelet count greater than or equal to 100 x 10^9/L.
9. Adequate renal function defined as:

   * Serum creatinine less than 1.5 mg/dL or calculated creatinine clearance greater than 50 mL/minute per the Cockcroft-Gault formula 10 Adequate liver function defined as:
   * Total Bilirubin within normal limits
   * Alkaline phosphatase (AP), alanine transaminase (ALT), and aspartate transaminase (AST) less than or equal to 2.5 x upper limit of normal (ULN)
   * AP, ALT, and AST less than or equal to 5 x ULN in the case of liver metastases and liver-specific AP less than or equal to 3 x ULN in the case of bone metastases 11 Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1.

12. Life expectancy greater than 3 months.

Exclusion Criteria:

Subjects who meet any of the following criteria are not eligible to participate in this study:

1. Known human immunodeficiency virus (HIV), clinical evidence of active viral hepatitis B or C, or severe/uncontrolled infections or intercurrent illness that is unrelated to the tumor.
2. Prior surgery, radiotherapy, chemotherapy, biologic therapy, or investigational agents within 4 weeks prior to the first infusion and prior immunotherapy, hormonal, or molecular-targeted therapy within 2 weeks prior to the first infusion. All acute toxicities related to prior treatments should have resolved.
3. Active malignancy other than the present diagnosis within the past 24 months (except treated non-melanoma skin cancer or carcinoma in situ of the cervix).
4. QT interval corrected for rate (QTc) greater than 450 msec on the electrocardiogram (ECG) obtained at Screening (Day -21 to 0) using the Fridericia method for QTc analysis.
5. History or substance or alcohol abuse which, in the opinion of the investigator, would prohibit participation in the study.
6. History of clinically significant cardiac impairment, congestive heart failure, New York Heart Association (NYHA) cardiac disease classification Class II, unstable angina, or myocardial infarction during the previous 6 months, or serious cardiac arrhythmia.
7. Current significant co-morbid disease which, in the opinion of the investigator, would exclude the subject from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-06-22 (Actual); Primary Completion 2011-08-01 (Actual); Study Completion 2015-10-15 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and dose-limiting toxicities as determined in Part A. | During Cycle 1: 28 days
Safety parameters (adverse events, laboratory data, vital signs, electrocardiogram data, Eastern Cooperative Oncology Group [ECOG] scores, and physical and neurological exams). | During Parts A and B: approximately 26 months

SECONDARY OUTCOMES:
Pharmacokinetics | Obtained prior to infusion on Day 1 of Cycle 1 (Baseline), during the infusion at 15 and 30 minutes (just prior to end of infusion), then after the end of infusion at 5 and 30 minutes, and 1, 2, 4, 8, 24, and 48 hours on Days 1 and 15 of Cycle 1 only.
Pharmacodynamics | Prior to and post-infusion at timepoints between Days 1 and 15, and on Day 1 of Cycle 2
Preliminary efficacy: Tumor assessments of objective response rate based on review of computed tomography and magnetic resonance imaging scans using Modified Response Evaluation Criteria in Solid Tumors. | Performed at baseline and every other cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Eisai Medical Services, Study Director — Eisai Inc.
Locations (12):
- United States (12):
  - Scottsdale, Arizona
  - Los Angeles, California
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Albany, New York
  - Greenville, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Norfolk, Virginia
  - Vancouver, Washington